CLINICAL TRIAL: NCT04991818
Title: Evaluating the User Experience of the OneBiome Consumers Value Journey Service Offered to the 1000 Days and Young Children Consumers Market
Brief Title: MSC - OneBiome UX Pilot Study
Acronym: OneBiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Chiang Children's Allergy and Asthma Clinic (Unknown); The Child and Allergic Clinic (Unknown); KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SBB20R&33310
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Microbial Colonization
Keywords: OneBiome; Consumer insights; User experience
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women or children 0-5 years of age (Experimental): Pregnant women in third trimester or children 0-5 years of age
  Interventions: Other: OneBiome microbiome profiling service

INTERVENTIONS:
Other: OneBiome microbiome profiling service — participants will be asked to complete the user experience of the OneBiome service

SUMMARY:
Evaluating the user (pregnant women and parents of young children) experience of the OneBiome consumers value journey service offered to the 1000 days and young children consumers market

DETAILED DESCRIPTION:
The OneBiome service aims to empower consumers with microbiome science in a friendly/consumer centric manner. The investigators wants to show that microbiome data can be used as an estimate of consumer's health and can be translated into actionable insights. The investigators aim to pilot a consumers' insight study to measure the perception/sentiments of this service in the Singapore market by recruiting study subjects from local public/private hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who are in the third trimester, or children from birth to 5 years of age
2. Pregnant women or parents of children should have access to the internet and a smartphone or tablet to access the OneBiome mobile friendly website.
3. Pregnant women or parents of children should be able to comprehend the content in the OneBiome mobile friendly website and complete the questionnaires in English.
4. Pregnant women and parents of children should stay in Singapore and remain contactable should they decide to do two microbiome assessments within 8 weeks

Exclusion Criteria:

1. Children born prematurely
2. Incapability of the pregnant women or parents of children to access OneBiome mobile friendly website and complete the questionnaires in English.
3. Any other family member is enrolled in the study
4. Incapability of the pregnant women or parents of children to comply with study protocol or Investigator's uncertainty about the willingness or ability of the pregnant women or parents of children to comply with the protocol requirements

Min Age: 0 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Overall user experience of the OneBiome microbiome profiling service | Approximately 8 weeks
  Pregnant women and parents of young children reported overall user experience of the OneBiome microbiome profiling service, i.e. average rating of the four following UX surveys1) overall experience of kit discovery (from unboxing to shipment); 2) ease of use of the stool collection kit; 3) overall user experience of the OneBiome web platform; 4) overall user experience of reading and understanding the microbiome analysis report.

SECONDARY OUTCOMES:
User experience of different "steps/ phases" of the OneBiome consumers value journey service | Approximately 8 weeks
  Pregnant women and parents of young children reported user experience of different "steps/ phases" of the OneBiome consumers value journey service, including 'kit discovery, 'kit usage', 'web platform', 'evaluation of report', 'evaluation of service' and ''evaluation of consumer's motivation and consumption behaviour habits'
Healthcare professional (HCP) reported overall experience of the OneBiome consumers value journey service | Approximately 8 weeks
  HCP reported overall user experience of the OneBiome microbiome profiling service
HCP reported usefulness of microbiome data | Approximately 8 weeks
  HCP reported usefulness of microbiome data for their general practice based on user experience interaction between HCP and pregnant women and parents of young children

OTHER OUTCOMES:
Microbiome composition of the participants | Approximately 8 weeks
  Microbiome composition in the stool sample of the subject which will be included in the microbiome analysis report to be shared with subject/ parent's subject.
Association between microbiome composition and known factors that influence the microbiome | Approximately 8 weeks
  Association between microbiome composition and known factors that influence the microbiome in early life including mode of delivery, antibiotic prophylaxis, infant feeding patterns and diet.
Food frequency questionnaire translation into food groups | Approximately 8 weeks
  FFQ data at the beginning and at the end of the study based on translation of FFQ into food groups according to the healthy plate guideline from the Health Promotion Board.
Association between gut health parameters, stool images, microbiome composition and dietary patterns | Approximately 8 weeks
  Association between gut health parameters (symptoms, stool consistency, frequency and color, gastrointestinal infection, antibiotic intake) and stool images from participants, and microbiome composition and dietary patterns

CONTACTS AND LOCATIONS:
Overall Officials: Bee Wah Lee, MD, Principal Investigator — The Child and Allergy Clinic; Wen Chin Chiang, MD, Principal Investigator — Chiang Children's Allergy and Asthma Clinic; Anne Goh, MD, Principal Investigator — KK Women's and Children's Hospital
Locations (2):
- Singapore (2):
  - Mount Elizabeth Medical Centre, Singapore
  - KK Women's and Children's Hospital, Singapore